CLINICAL TRIAL: NCT07105293
Title: Effects of Different Peep Applications on Tissue Oxygenation, Respiratory Mechanics and Postoperative Pulmonary Complications in Laparoscopic Hysterectomy Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Büşra Şabano, Research Assistant, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBU-AVR-BS-01
Record Dates: First submitted 2025-06-25; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Laparoscopy; Positive End Expiratory Pressure (PEEP); Respiratory Mechanics
Keywords: Laparoscopic hysterectomy; PEEP; Postoperative pulmonary complications; Respiratory mechanics; Driving pressure; Tissue oxygenation

STUDY DESIGN:
Intervention Model Description: Patients were randomized into two equal groups; one group received PEEP 5 cmH₂O, while the other received PEEP 10 cmH₂O.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEP 5 cmH2o applied group (Active Comparator): A standardized anesthesia protocol involved volume-controlled ventilation with a tidal volume of 6-8 mL/kg and a frequency of 10-12 breaths/min. Patients were randomized into two equal groups; one group received PEEP 5 cmH₂O
  Interventions: Other: PEEP 5 cmH2o applied group
- PEEP 10 cmH2o applied group (Active Comparator): A standardized anesthesia protocol involved volume-controlled ventilation with a tidal volume of 6-8 mL/kg and a frequency of 10-12 breaths/min. Patients were randomized into two equal groups; one group received PEEP 10 cmH₂O
  Interventions: Other: PEEP 10 cmH2o applied group

INTERVENTIONS:
Other: PEEP 5 cmH2o applied group — A standardized anesthesia protocol involved volume-controlled ventilation with a tidal volume of 6-8 mL/kg and a frequency of 10-12 breaths/min, PEEP:5 cmH2o
  Arms: PEEP 5 cmH2o applied group
Other: PEEP 10 cmH2o applied group — A standardized anesthesia protocol involved volume-controlled ventilation with a tidal volume of 6-8 mL/kg and a frequency of 10-12 breaths/min, PEEP:10 cmH2o
  Arms: PEEP 10 cmH2o applied group

SUMMARY:
This study aims to compare the effects of two different PEEP levels (5 cmH₂O and 10 cmH₂O) during laparoscopic hysterectomy on perioperative tissue and cerebral oxygenation, respiratory mechanics, and postoperative pulmonary complications.

DETAILED DESCRIPTION:
Laparoscopic surgery is frequently performed today due to its rapid recovery, short hospital stay, minimal incisions, and minimal postoperative pain. Despite these advantages of laparoscopic hysterectomy, the patient's Trendelenburg position and pneumoperitoneum can cause abdominal organs to shift to the diaphragm, decrease lung compliance, atelectasis, and ultimately compromise respiratory function and mechanics. Tissue hypoxia occurs, affecting cerebral perfusion. Consequently, these patients are prone to perioperative hypoxemia and postoperative pulmonary complications. PEEP can improve arterial oxygenation and reduce atelectasis. The aim of this study was to compare the effectiveness of PEEP in terms of perioperative tissue oxygenation, cerebral perfusion, respiratory mechanics, and postoperative pulmonary complications.

The study was planned to include 64 patients aged 18-75 years, with ASA status I-III, who provided informed consent and were undergoing elective laparoscopic hysterectomy. The patients were randomized into two groups: one with PEEP 5 cmH₂O and the other with PEEP 10 cmH₂O. The aim was to compare the two groups' hemodynamic variables, NIRS values, peak inspiratory pressure (Ppeak), plateau pressure (Pplato), mean airway pressure (Pmean), end-tidal CO₂ (EtCO₂), driving pressure, serum lactate, partial arterial oxygen (PaO2), and carbon dioxide (PaCO2) levels, recorded after intubation, 30 minutes after pneumoperitoneum, and 15 minutes after desufflation. The ARISCAT score was used to assess the risk of any postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* The study group included patients aged 18-70 years with ASA physical status I-III who were scheduled for elective laparoscopic hysterectomy under general anesthesia between November 1, 2023 and February 15, 2024 and who gave informed consent for participation.

Exclusion Criteria:

* Previous history of pneumothorax
* ASA IV classification
* Significant pulmonary impairment (moderate/severe chronic obstructive pulmonary disease, emphysema, pulmonary hypertension, etc.)
* Active upper respiratory tract infection or recurrent respiratory infections requiring recent antibiotic treatment
* Severe systemic diseases
* Heavy smoking (≥20 pack-years)
* Emergency surgical cases
* Failure to provide written informed consent for any reason
* Contraindications to PEEP application

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Intergroup comparison of near infrared spektroscopy (NIRS) value | During the operation
  Comparison of near infrared spektroscopy (NIRS) values between two groups with PEEP: 5 mmHg and PEEP: 10 mmHg baseline, after intubation, after pneumoperitoneum and after insufflation
Pulmonary Outcomes | During the operation
  It was determined whether pulmonary complications developed and its relationship with the Ariscat score was evaluated.
  Ariscat score:
  Low Risk: 0-26 point Middle Risk: 26-44 point Hihg Risk: 45≤ point
Intergroup comparison of peak inspiratory pressure (Ppeak) value (mmHg) | During the operation
  Comparison of peak inspiratory pressure (Ppeak) values between two groups with PEEP: 5 mmHg and PEEP: 10 mmHg after intubation, after pneumoperitoneum and after insufflation
Intergroup comparison of plato pressure (Ppeak) value (mmhg) | during the operation
  Comparison of plato pressure (Pplato) values between two groups with PEEP: 5 mmHg and PEEP: 10 mmHg after intubation, after pneumoperitoneum and after insufflation
Intergroup comparison of mean airway pressure (Pmean) value (mmhg) | during the operation
  Comparison of mean airway pressure (Pmean) values between two groups with PEEP: 5 mmHg and PEEP: 10 mmHg after intubation, after pneumoperitoneum and after insufflation
Intergroup comparison of end tidal carbondioxide (EtCO2) value (mmhg) | during the operations
  Comparison of end tidal carbondioxide (EtCO2) values between two groups with PEEP: 5 mmHg and PEEP: 10 mmHg after intubation, after pneumoperitoneum and after insufflation
Intergroup comparison of driving pressure value (mmhg) | during the operations
  Comparison of driving pressure values between two groups with PEEP: 5 mmHg and PEEP: 10 mmHg after intubation, after pneumoperitoneum and after insufflation
Intergroup comparison of partial oxygen pressures (PaO2) (mmhg) | during the operations
  Comparison of partial oxygen pressures (pao2) in arterial blood gas between two groups with PEEP: 5 mmHg and PEEP: 10 mmHg after intubation, after pneumoperitoneum and after insufflation
Intergroup comparison of partial carbondioxide pressures (PaCO2) (mmhg) | during the operations
  Comparison of partial carbondioxide pressures (PaCO2) in arterial blood gas between two groups with PEEP: 5 mmHg and PEEP: 10 mmHg after intubation, after pneumoperitoneum and after insufflation
Intergroup comparison of lactate value | during the operation
  Comparison of lactate values between two groups with PEEP: 5 mmHg and PEEP: 10 mmHg after intubation, after pneumoperitoneum and after insufflation

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr. Lutfi Kirdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No